CLINICAL TRIAL: NCT04021862
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Bermekimab in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of Bermekimab in Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108833; 77474462ADM2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm 1 (bermekimab every week) (Experimental): Loading Dose: 400 mg subcutaneous (SC) injection of bermekimab and a SC injection of matching placebo at week 0 (Baseline).
  Treatment Dose: 400 mg subcutaneous injection of bermekimab administered weekly (qw) from week 1 through Week 31.
  Interventions: Drug: Bermekimab Monoclonal Antibody; Drug: Placebo
- Treatment Arm 2 (bermekimab every other week) (Experimental): Loading Dose: 800 mg SC injection of bermekimab at week 0 (Baseline).
  Treatment Dose: 400 mg SC injection of bermekimab administered every other week (q2w) alternating with matching placebo q2w through Week 31.
  Interventions: Drug: Bermekimab Monoclonal Antibody; Drug: Placebo
- Placebo (Placebo Comparator): Loading Dose: Placebo matching to bermekimab (4 milliliters [mL]) SC injection at Week 0, (Baseline).
  Treatment Dose: SC injection of matching placebo administered once weekly (qw) from week 1 to week 15 during placebo-controlled period. After completion of placebo-controlled period, participants will cross-over and receive bermekimab 400 mg SC injection qw at Week 16 through Week 31.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bermekimab Monoclonal Antibody — Bermekimab 400 mg or 800 mg will be administered subcutaneously.
  Arms: Treatment Arm 1 (bermekimab every week); Treatment Arm 2 (bermekimab every other week)
Drug: Placebo — Placebo will be administered subcutaneously.

SUMMARY:
A Study to Evaluate the Safety and Efficacy of Bermekimab in Patients With Moderate to Severe Atopic Dermatitis

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blind, placebo-controlled study of bermekimab in patients with moderate to severe atopic dermatitis. The primary objective of the study is to analyze the safety and efficacy of different dose regimens of bermekimab compared to placebo treatment in adult patients with moderate-to-severe AD. The study is multicenter and will consist of three groups:

Treatment Arm 1: Bermekimab every week (qw)

Treatment Arm 2: Bermekimab every other week (q2w)

Arm 3 (Placebo): Placebo every week (qw)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years
* Willing and able to attend all clinic visits and comply with study-related procedures
* Participant can understand and complete study-related questionnaires
* Written informed consent provided by the participant
* Chronic atopic dermatitis present for at least 3 years
* Eczema Area and Severity Index Score (EASI) score greater than or equal to (>=) 16 at screening and baseline visits
* Investigators Global Assessment (IGA) >= 3 at screening and baseline visits
* Baseline pruritis numerical rating scale average score for maximum intensity of at least 3, based on the average of daily pruritis numerical rating scale scores for maximum itch intensity reported during the 7 days prior to randomization
* Has applied a stable dose of topical moisturizer twice daily for at least 7 consecutive days immediately prior to the baseline visit and is willing to continue this regimen on a daily basis for the duration of the study
* >= 10 percent (%) body surface area (BSA) of Atopic Dermatitis (AD) involvement at screening and baseline visits
* Documented recent history (within 6 months prior to screening) of inadequate response to treatment with topical medications, or participants for whom topical treatments are medically inadvisable (because of important side effects or safety risks): (a) Inadequate response is defined as failure to achieve and maintain remission or a low disease activity state (comparable to an IGA score of 0-2), despite treatment with a daily regimen of topical corticosteroids of medium to higher potency (with or without topical calcineurin inhibitors as appropriate), applied for at least 28 days or for the maximum duration recommended by the product prescribing information, whichever is shorter; (b) Participants with documented systemic treatment for atopic dermatitis in the preceding 6 months are also considered to be inadequate responders to topical treatments and are potentially eligible for treatment with MABp1, after appropriate washout; (c) Important side effects or risks are those that outweigh the potential treatment benefits, and include: intolerance to treatment, hypersensitivity reactions, significant skin atrophy, and adverse systemic effects; and (d) Acceptable documentation includes contemporaneous chart notes that record topical medication prescription and treatment outcome, or investigator documentation based on communication with the participant's treating physician.

Exclusion Criteria:

* Participants has been treated for AD with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) of the drug prior to baseline
* Treatment with bermekimab at any time in the past
* Treatment with immunosuppressive/immunomodulatory drugs or phototherapy for atopic dermatitis within 4 weeks of baseline, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment
* Treatment with topical corticosteroids or topical calcineurin inhibitors for the treatment of AD within 14 days prior to baseline
* Treatment with biologics as follows: (a) Any cell-depleting agents including, but not limited to, rituximab, within 5 half-lives (if known) or 30 days prior to baseline visit, or until lymphocyte count returns to normal, whichever is longer; (b) Other biologics: within 5 half-lives (if known) or 30 days prior to baseline visit, whichever is longer
* Initiation of treatment of atopic dermatitis with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (participants may continue to use stable doses of such moisturizers if initiated before the screening visit)
* Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit
* Planned or anticipated use of any prohibited medications and procedures during study treatment
* Treatment with a live (attenuated) vaccine within 30 days prior to the screening visit
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to the baseline visit, or superficial skin infections within 1 week prior to the baseline visit
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (for example, tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis, aspergillosis) despite infection resolution; or unusually frequent, recurrent, or prolonged infections, per investigator judgment
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening
* Positive for hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody at the screening visit
* At baseline, presence of any conditions listed as criteria for study drug discontinuation
* Presence of skin comorbidities that may interfere with study assessments
* History of malignancy within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, and completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin diagnosed active endoparasitic infections; suspected or high risk of endoparasitic, unless clinical and (if necessary) laboratory assessments have ruled out active infection before randomization
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the Participant's participation in the study. Examples include, but are not limited to, participants with short life expectancy, participants with uncontrolled diabetes (HbA1c >= 9%), participants with cardiovascular conditions (for example, stage III or IV cardiac failure according to the New York Heart Association classification), severe renal conditions (for example, participants on dialysis), hepato-biliary conditions (for example, Child-Pugh class B or C), neurological conditions (for example, demyelinating diseases), active major autoimmune diseases (for example, lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), other severe endocrinological, gastrointestinal, metabolic, pulmonary or lymphatic diseases. The specific justification for participants excluded under this criterion will be noted in study documents (chart notes, case report forms [CRFs], etc.)
* Planned or anticipated major surgical procedure during the participant's participation in this study
* Membership of the investigational team or his/her immediate family
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study
* Women unwilling to use adequate birth control, if of reproductive potential and sexually active. Adequate birth control is defined as consistent practice of an effective and accepted method of contraception throughout the duration of the study and for 120 days after the last dose of study drug. These methods include hormonal contraceptives, intrauterine device, double barrier contraception (that is, condom + diaphragm), or male partner with a documented vasectomy
* History of severe allergic or anaphylactic reactions to monoclonal antibodies
* Any other medical or psychological condition (including relevant laboratory abnormalities at screening) that, in the opinion the investigator, may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study participant as a result of his/her participation in the study, may make participant's participation unreliable, or may interfere with study assessments. The specific justification for participant excluded under this criterion will be noted in study documents (chart notes, case report forms, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (17):
  - Beach Clinical Research Inc, Huntington Beach, California
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Doral Medical Research, Doral, Florida
  - Floridian Research Institute, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - Premier Research Associate, Inc, Miami, Florida
  - CNS HealthCare, Orlando, Florida
  - Avita Clinical Research, Tampa, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Randall Dermatology & Cosmetic Surgery, West Lafayette, Indiana
  - Revival Research Institute LLC, Troy, Michigan
  - ClinOhio Research Services, Columbus, Ohio
  - Helios Clinical Research, LLC, Milan, Tennessee
  - Progressive Clinical Research, San Antonio, Texas
  - Dominion Medical Associates, Inc., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Week 0 - 16): Participants received placebo matching to bermekimab (4 milliliters [mL]) subcutaneous (SC) injection at Week 0, followed by weekly (qw) placebo SC injections from Week 1 through Week 16.
- Bermekimab 400 mg q2w (Week 0 - 16): Participants received bermekimab 800 milligrams (mg) (400mg*2) loading dose SC injection at Week 0 followed by bermekimab 400 mg SC injections every 2 weeks (q2w) alternating with matching placebo q2w through Week 16.
- Bermekimab 400 mg qw (Week 0 - 16): Participants received bermekimab 400 mg loading dose SC injection along with matching placebo loading dose SC injection at Week 0 followed by weekly (qw) SC injections of bermekimab 400 mg (2*200 mg per mL) through Week 16.
- Placebo Then Bermekimab 400 mg qw (Week 16 - 31): After completion of placebo-controlled period, participants were crossed-over to active treatment period and received bermekimab 400 mg SC injection qw at Week 16 through Week 31.
- Bermekimab 400 mg q2w (Week 16 - 31): After completion of placebo-controlled period, participants entered active treatment period and continued to receive bermekimab 400 mg SC injection q2w alternating with matching placebo through Week 31.
- Bermekimab 400 mg qw (Week 16 - 31): After completion of placebo-controlled period, participants entered active treatment period and continued to receive bermekimab 400 mg SC injection qw through Week 31.
Period: Placebo Controlled Period (Week 0-16)
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Started | 29 | 29 | 29 | 0 | 0 | 0
Completed | 27 | 28 | 27 | 0 | 0 | 0
Not Completed | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0
Period: Active Treatment Period (Week 16-32)
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Started | 0 | 0 | 0 | 27 | 28 | 27
Completed | 0 | 0 | 0 | 26 | 28 | 27
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Total
Number analyzed (Participants) | 29 | 29 | 29 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (15.59) | 44 (15.71) | 41.9 (16.65) | 45.5 (16.25)
Age, Customized [Number; unit: participants]
  Adults (18-64 years) | 23 | 27 | 27 | 77
  From 65 to 84 years | 5 | 2 | 2 | 9
  85 years and over | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 20 | 58
  Male | 9 | 11 | 9 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 8 | 22
  White | 23 | 19 | 20 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 29 | 29 | 29 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index-75 (EASI-75) Response at Week 16
Description: Percentage of participants achieving EASI-75 at Week 16 were reported. EASI-75 response was defined as at least 75% improvement from baseline in EASI total score. The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The total EASI score is the sum of four body-region scores ranged from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16)
Number analyzed (Participants) | 29 | 29 | 29
percentage of participants | 13.8 | 24.1 | 34.5

2. Secondary Outcome: Percentage of Participants Achieving >=4 Point Improvement (Reduction From Baseline) in Weekly Average Peak (Worst) Daily Pruritus (Itch) Numeric Rating Scale (NRS) Score From Baseline at Week 4, 8, 12, 16 and 32 Among Participants With Baseline Score >=4
Description: Percentage of participants achieving greater than or equal to (>=4) point improvement (reduction from baseline) in weekly average peak (worst) daily pruritus NRS score from baseline at Weeks 4, 8, 12, 16 and 32 among participants with a baseline score >=4 were reported. The eczema skin pain and itch NRS is a 2-item patient-reported outcome that participants used to rate the severity of their eczema-related skin pain and eczema related itch daily. To rate the severity of eczema-related itch participants were asked the following question: please rate the severity of your eczema-related itch at its worst in the past 24 hours. The response was rated on a 0 to 10 NRS ranging from 0 "none" to 10 "worst possible". Higher score indicated more severity. Seven daily average NRS scores are into a weekly score.
Time Frame: Weeks 4, 8, 12, 16 and 32
Population: FAS included all randomized participants who received at least 1 dose of study agent. Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure, n (number analyzed) signifies number of participants who were analyzed at the specified timepoints and '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 26 | 25 | 23 | 25 | 25 | 23
percentage of participants
  Week 4: number analyzed (Participants) | 26 | 25 | 23 | 0 | 0 | 0
  Week 4 | 26.9 | 8.0 | 8.7 |  |  |
  Week 8: number analyzed (Participants) | 26 | 25 | 23 | 0 | 0 | 0
  Week 8 | 34.6 | 16.0 | 26.1 |  |  |
  Week 12: number analyzed (Participants) | 26 | 25 | 23 | 0 | 0 | 0
  Week 12 | 46.2 | 28.0 | 30.4 |  |  |
  Week 16 | 53.8 | 32.0 | 52.2 | 56.0 | 32.0 | 52.2
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 25 | 25 | 23
  Week 32 |  |  |  | 80.0 | 64.0 | 65.2

3. Secondary Outcome: Percentage of Participants Achieving >= 4 Point Improvement (Reduction From Baseline) in Weekly Average of Average Daily Pruritis (Itch) NRS Score From Baseline at Weeks 4, 8, 12, 16 and 32 Among Participants With a Baseline Score >=4
Description: Percentage of participants achieving >= 4 improvement (reduction from baseline) in weekly average of average daily pruritis NRS score from baseline at Weeks 4, 8, 12, 16 and 32 among participants with a baseline score >=4 were reported. The eczema skin pain and itch NRS is a 2-item patient-reported outcome that participants used to rate the severity of their eczema-related skin pain and eczema related itch daily. To rate the severity of eczema-related itch participants were asked the following question: please rate the severity of your eczema-related average itch in the past 24 hours. The response was rated on a 0 to 10 NRS. Higher score indicated more severity. Seven daily averaged NRS scores were averaged into a weekly score.
Time Frame: Weeks 4, 8, 12, 16 and 32
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 26 | 22 | 22 | 14 | 12 | 17
percentage of participants
  Week 4: number analyzed (Participants) | 26 | 22 | 22 | 0 | 0 | 0
  Week 4 | 23.1 | 13.6 | 9.1 |  |  |
  Week 8: number analyzed (Participants) | 26 | 22 | 22 | 0 | 0 | 0
  Week 8 | 30.8 | 22.7 | 27.3 |  |  |
  Week 12: number analyzed (Participants) | 26 | 22 | 22 | 0 | 0 | 0
  Week 12 | 50.0 | 27.3 | 40.9 |  |  |
  Week 16 | 50.0 | 50.0 | 54.5 | 35.7 | 25.0 | 47.1
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 14 | 12 | 17
  Week 32 |  |  |  | 71.4 | 66.7 | 58.8

4. Secondary Outcome: Percentage of Participants Achieving >=4 Improvement (Reduction From Baseline) in Weekly Average Peak (Worst) Daily Skin Pain NRS Score From Baseline at Weeks 4, 8, 12, 16 and 32 Among Participants With a Baseline Score >=4
Description: Percentage of participants achieving >=4 improvement (reduction from baseline) in weekly average peak (worst) daily skin pain NRS score from baseline at Weeks 4, 8, 12, 16 and 32 among participants with a baseline score >=4 were reported. The eczema skin pain and Itch NRS is a 2-item patient-reported outcome that participants used to rate the severity of their eczema-related skin pain and eczema related itch daily. To rate the severity of eczema-related skin pain participants were asked the following question: Please rate the severity of your eczema-related skin pain at its worst in the past 24 hours. The response was rated on a 0 to 10 NRS ranging from 0 "none" to 10 "worst possible". Seven daily NRS scores were averaged into a weekly score. Higher score indicated more severity.
Time Frame: Weeks 4, 8, 12, 16 and 32
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 17 | 17 | 20 | 16 | 17 | 20
percentage of participants
  Week 4: number analyzed (Participants) | 17 | 17 | 20 | 0 | 0 | 0
  Week 4 | 47.1 | 23.5 | 25.0 |  |  |
  Week 8: number analyzed (Participants) | 17 | 17 | 20 | 0 | 0 | 0
  Week 8 | 41.2 | 29.4 | 30.0 |  |  |
  Week 12: number analyzed (Participants) | 17 | 17 | 20 | 0 | 0 | 0
  Week 12 | 41.2 | 17.6 | 40.0 |  |  |
  Week 16 | 35.3 | 29.4 | 40.0 | 37.5 | 29.4 | 40.0
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 16 | 17 | 20
  Week 32 |  |  |  | 56.3 | 52.9 | 50.0

5. Secondary Outcome: Percentage of Participants Achieving >=4 Improvement (Reduction From Baseline) in Weekly Average of Average Daily Skin Pain NRS Score From Baseline at Weeks 4, 8, 12, 16 and 32 Among Participants With a Baseline Score >=4
Description: Percentage of participants achieving >=4 improvement (reduction from baseline) in weekly average of average daily skin pain NRS score from baseline to Weeks 4, 8, 12, 16 and 32 among participants with a baseline score >=4 were reported. The eczema skin pain and Itch NRS is a 2-item patient-reported outcome that participants used to rate the severity of their eczema-related skin pain and eczema related itch daily. To rate the severity of eczema-related skin pain participants were asked the following question: Please rate the severity of your eczema-related average skin pain in the past 24 hours; The response was rated on a 0 to 10 NRS. Higher score indicated more severity. Seven daily averaged NRS scores were averaged into a weekly score.
Time Frame: Weeks 4, 8, 12, 16 and 32
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 15 | 12 | 17 | 14 | 12 | 17
percentage of participants
  Week 4: number analyzed (Participants) | 15 | 12 | 17 | 0 | 0 | 0
  Week 4 | 40.0 | 33.3 | 17.6 |  |  |
  Week 8: number analyzed (Participants) | 15 | 12 | 17 | 0 | 0 | 0
  Week 8 | 33.3 | 50.0 | 35.3 |  |  |
  Week 12: number analyzed (Participants) | 15 | 12 | 17 | 0 | 0 | 0
  Week 12 | 40.0 | 33.3 | 52.9 |  |  |
  Week 16 | 33.3 | 25.0 | 47.1 | 35.7 | 25.0 | 47.1
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 14 | 12 | 17
  Week 32 |  |  |  | 71.4 | 66.7 | 58.8

6. Secondary Outcome: Percentage of Participants Achieving EASI-75 Response at Weeks 4, 8, 12, and 32
Description: Percentage of participants achieving EASI-75 response at Weeks 4, 8, 12, and 32 were reported. EASI-75 response was defined as at least 75% improvement from baseline in EASI total score. The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The total EASI score is the sum of four body-region scores ranged from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Weeks 4, 8, 12, and 32
Population: FAS included all randomized participants who received at least 1 dose of study agent. Here, n (number analyzed) signifies number of participants who were analyzed at the specified timepoints and '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 28 | 27
percentage of participants
  Week 4: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 4 | 10.3 | 17.2 | 10.3 |  |  |
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | 10.3 | 13.8 | 17.2 |  |  |
  Week 12: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 12 | 13.8 | 20.7 | 37.9 |  |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 28 | 27
  Week 32 |  |  |  | 77.8 | 69.0 | 65.5

7. Secondary Outcome: Percentage of Participants With an Investigators Global Assessment (IGA) Score of 0 or 1 and a Reduction From Baseline of >=2 Points at Week 16
Description: Percentage of participants with both IGA score of 0 or 1 and a reduction from baseline of >=2 points was reported. IGA assesses AD severity and clinical response using a 5-point scale: 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, 4 = severe. A higher score indicated more severity of AD. The score was determined by ranking the extent of erythema and population/infiltration. A clinical response to therapy was an IGA score of 0 (clear) or 1 (almost clear). This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16)
Number analyzed (Participants) | 29 | 29 | 29
percentage of participants
  IGA score of clear (0) | 0 | 6.9 | 6.9
  IGA score of clear (0) or almost clear (1) | 6.9 | 17.2 | 13.8
  IGA score of mild or better (reduction from baseline of >=2 points) | 24.1 | 34.5 | 34.5

8. Secondary Outcome: Percentage of Participants Achieving EASI-90 Response at Weeks 12, 16, and 32
Description: Percentage of participants achieving EASI-90 response at Weeks 12, 16 and 32 were reported. EASI-90 response was defined as at least 90% improvement from baseline in EASI total score. The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The total EASI score is the sum of four body-region scores ranged from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Weeks 12, 16, and 32
Population: FAS; N (number of participants analyzed)=participants evaluated for this outcome measure, n (number analyzed)=participants analyzed at specified timepoints, 0=no participant analyzed. Week 16 data were collected and analyzed only for placebo crossover participants during active treatment period as pre-planned. For active treatment period assessments, participants who discontinued placebo controlled period in Bermekimab 400 mg q2w and Bermekimab 400 mg qw arms were also included as pre-planned.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
percentage of participants
  Week 12: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 12 | 6.9 | 6.9 | 10.3 |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | 0 | 10.3 | 10.3 | 0 |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | 37.0 | 24.1 | 34.5

9. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Weeks 8, 12, 16, and 32
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The format is a simple response (0 to 3 where 0 is "not at all" and 3 is "very much") to 10 questions, which assess QOL over the past week, with an overall scoring system of 0 to 30. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. A higher score indicates more severe disease and poor QoL.
Time Frame: Baseline, Weeks 8, 12, 16 and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
score on a scale
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | -4.86 (5.598) | -3.03 (4.136) | -3.41 (4.694) |  |  |
  Week 12: number analyzed (Participants) | 29 | 28 | 29 | 0 | 0 | 0
  Week 12 | -4.86 (5.774) | -3.29 (3.505) | -4.72 (5.028) |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | -6.07 (7.151) | -3.38 (3.886) | -5.93 (5.120) | -6.52 (7.213) |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | -9.15 (6.413) | -4.10 (5.759) | -7.76 (6.122)

10. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) (Anxiety) Score at Weeks 8, 12, 16, and 32
Description: In this outcome measure, change from baseline in HADS-Anxiety score at weeks 8, 12, 16 and 32 were reported. The HADS is an instrument for screening anxiety and depression in non-psychiatric populations; repeated administration also provides information about changes to a participant's emotional state. The HADS is a 14-item self-administered questionnaire, 7 each for anxiety and depression symptoms. Each item is scored from 0-3, resulting in total anxiety score ranging from 0 (less severity of anxiety) to 21 (greater severity of anxiety). Higher score indicated more anxiety symptoms. The following cut-off scores are recommended: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety.
Time Frame: Baseline, Weeks 8,12,16 and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
score on a scale
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | 1.59 (2.732) | 2.00 (3.770) | 1.90 (2.257) |  |  |
  Week 12: number analyzed (Participants) | 29 | 28 | 29 | 0 | 0 | 0
  Week 12 | 1.45 (2.898) | 1.89 (3.755) | 2.62 (2.846) |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | 1.59 (2.771) | 1.97 (3.669) | 2.66 (3.062) | 1.70 (2.839) |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | 2.93 (3.419) | 2.34 (3.467) | 3.14 (3.114)

11. Secondary Outcome: Change From Baseline in HADS (Depression) Score at Weeks 8, 12, 16, and 32
Description: In this outcome measure, change from baseline in HADS-depression score at weeks 8, 12, 16 and 32 were reported. The HADS is an instrument for screening anxiety and depression in non-psychiatric populations; repeated administration also provides information about changes to a participant's emotional state. The HADS is a 14-item self-administered questionnaire, and consists of 7 items each for anxiety and depression symptoms. Each item is scored from 0-3, resulting in total depression score ranging from 0 (less severity of depression) to 21 (greater severity of depression). Higher score indicated more depression symptoms. The following cut-off scores are recommended: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe depression.
Time Frame: Baseline, Weeks 8,12,16 and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
score on a scale
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | 0.86 (1.941) | 0.59 (3.088) | 1.31 (2.904) |  |  |
  Week 12: number analyzed (Participants) | 29 | 28 | 29 | 0 | 0 | 0
  Week 12 | 0.97 (2.291) | 0.57 (3.132) | 0.90 (3.426) |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | 0.93 (2.103) | 0.31 (2.989) | 1.07 (3.139) | 1.00 (2.166) |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | 1.93 (2.235) | 0.28 (3.401) | 1.55 (4.188)

12. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Scores at Weeks 8, 12, 16, and 32
Description: The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults. Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema). Higher scores indicated more severe disease and poor quality of life.
Time Frame: Baseline, Weeks 8, 12, 16, and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
score on a scale
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | -4.79 (3.949) | -5.66 (5.627) | -6.59 (4.939) |  |  |
  Week 12: number analyzed (Participants) | 29 | 28 | 29 | 0 | 0 | 0
  Week 12 | -5.07 (5.021) | -6.14 (5.543) | -7.55 (4.903) |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | -5.76 (5.680) | -6.00 (5.542) | -8.07 (5.618) | -6.19 (5.657) |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | -10.48 (6.659) | -8.66 (6.726) | -10.66 (6.800)

13. Secondary Outcome: Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Total Score at Weeks 8, 12, 16, and 32.
Description: SCORAD is a validated scoring index for AD, which consists of 3 components that is A =extent or affected body surface area assessed as percentage of each defined body area and reported as the sum of all areas, with a maximum score of 100%. B=severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) assessed using the following scale: none (0), mild (1), moderate (2), or severe (3) (for a maximum of 18 total points) and C=subjective symptoms scored by participants on visual analogue scale, where "0" is no itch (or no sleeplessness) and "10" is worst imaginable itch (or sleeplessness) with a maximum score of 20. SCORAD total score was calculated using these 3 aspects: extent (A: 0-100), severity (B: 0-18), and subjective symptoms (C: 0-20) using the formula: A/5 + 7*B/2+ C to give the SCORAD total score range of 0 to 103, where 0 = no disease to 103 = severe disease. Higher values of SCORAD represent worse outcome.
Time Frame: Baseline to Weeks 8, 12, 16 and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
score on a scale
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | 21.53 (11.468) | 21.29 (15.632) | 19.39 (11.632) |  |  |
  Week 12: number analyzed (Participants) | 29 | 28 | 29 | 0 | 0 | 0
  Week 12 | 24.27 (13.130) | 26.50 (12.894) | 22.45 (12.849) |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | 25.90 (15.916) | 27.56 (13.661) | 24.11 (14.961) | 27.82 (14.743) |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | 44.35 (16.479) | 31.92 (18.467) | 35.05 (18.461)

14. Secondary Outcome: Change From Baseline in Global Individual Signs Score (GISS) at Weeks 8, 12, 16, and 32.
Description: GISS assesses AD lesions for erythema, excoriations, lichenification and edema/papulation. Each component was rated on a global basis (over the entire body surface rather than region) using a 4-point scale (0=none, 1=mild, 2=moderate and 3=severe) according to the EASI grading severity. The cumulative score, which ranges from 0 to 12, is the sum of the four components. A higher score indicates more severe disease.
Time Frame: Baseline, Weeks 8,12,16 and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 29 | 29
score on a scale
  Week 8: number analyzed (Participants) | 29 | 29 | 29 | 0 | 0 | 0
  Week 8 | 2.97 (1.973) | 3.24 (2.247) | 2.07 (2.034) |  |  |
  Week 12: number analyzed (Participants) | 29 | 28 | 29 | 0 | 0 | 0
  Week 12 | 3.48 (2.385) | 3.54 (2.516) | 2.93 (2.313) |  |  |
  Week 16: number analyzed (Participants) | 29 | 29 | 29 | 27 | 0 | 0
  Week 16 | 3.34 (2.768) | 3.69 (2.647) | 2.97 (2.514) | 3.59 (2.707) |  |
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 27 | 29 | 29
  Week 32 |  |  |  | 5.70 (2.799) | 3.97 (2.934) | 3.97 (2.860)

ADVERSE EVENTS:
Time Frame: Up to Week 36
Description: The safety analysis set included all randomized participants who received at least 1 (partial or complete) dose of study agent, that is, the treated population. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Arm/Group | Placebo (Week 0 - 16) | Bermekimab 400 mg q2w (Week 0 - 16) | Bermekimab 400 mg qw (Week 0 - 16) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) | Bermekimab 400 mg q2w (Week 16 - 31) | Bermekimab 400 mg qw (Week 16 - 31)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/27 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 1/29 | 0/27 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 2/29 | 7/29 | 2/29 | 3/27 | 3/28 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 - 16) (N=29) | Bermekimab 400 mg q2w (Week 0 - 16) (N=29) | Bermekimab 400 mg qw (Week 0 - 16) (N=29) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) (N=27) | Bermekimab 400 mg q2w (Week 16 - 31) (N=28) | Bermekimab 400 mg qw (Week 16 - 31) (N=27)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 - 16) (N=29) | Bermekimab 400 mg q2w (Week 0 - 16) (N=29) | Bermekimab 400 mg qw (Week 0 - 16) (N=29) | Placebo Then Bermekimab 400 mg qw (Week 16 - 31) (N=27) | Bermekimab 400 mg q2w (Week 16 - 31) (N=28) | Bermekimab 400 mg qw (Week 16 - 31) (N=27)
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 2 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The relatively small sample size combined with the heterogeneity of the atopic dermatitis (AD) population were considered limitations of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT04021862/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT04021862/SAP_001.pdf